CLINICAL TRIAL: NCT01992770
Title: STEP-UP - A Randomised Controlled Trial for the Study of a Stepped-care Model Including a Tailored Behavioural Medicine Pain Intervention in Primary Care
Brief Title: A Stepped-care Model of Tailored Behavioural Medicine Pain Intervention in Primary Care
Acronym: STEP-UP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organisational changes at primary care units.
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Rheumatism Ass (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/448
Record Dates: First submitted 2013-09-23; First posted 2013-11-25 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Musculoskeletal Pain
Keywords: behavioural medicine; pain; physical therapy; physical exercise; primary care
MeSH Terms: conditions — Musculoskeletal Pain; Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored behavioural medicine (Experimental): After having received a minimal intervention (step 1) comprising 'stay-active advice', participants scoring >90 on the Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) are randomly allocated to an eight-week treatment in step 2, depending on risk profile. The experimental condition includes supervised physical exercises integrated with either (a) graded activity, or (b) hierarchical graded exposure depending on risk profile, i.e. absence or presence of pain catastrophizing and fear-avoidance beliefs.
  Interventions: Behavioral: Hierarchical graded exposure; Behavioral: Graded activity; Behavioral: Physical exercises
- Control group (Active Comparator): Participants will be scheduled for supervised, regular Physical exercises twice a week during eight weeks 8. Participants with a "moderate to high disability" risk profile will receive: Tailored graded activities training.
  Interventions: Behavioral: Physical exercises

INTERVENTIONS:
Behavioral: Hierarchical graded exposure — Individual Behavioural goal identification, depending on risk profile
  (1a). "Catastrophising and/or fear-avoidance" (2); hierarchical graded exposure, organized with individual coaching in connection to the physical training sessions, based on activities that each participant fear and/or avoid.
  Arms: Tailored behavioural medicine
Behavioral: Graded activity — Individual Behavioural goal identification, depending on risk profile
  (1b) "Graded activity";(2) self-monitoring of everyday life activities (3) functional behavioural analyses to describe, predict, and verify factors controlling patient's current and future activity performance (4) training of motor skills, cognitive skills, and strategies to organise everyday life including social support. (5) gradual application of acquired skills in everyday life situations as formulated by Specific, Measureable, Activity-related, Realistic, and Time- specified (SMART) goal setting (6) generalisation of skills to additional activities and challenging situations, and (7) strategies for maintenance and relapse prevention.
  Arms: Tailored behavioural medicine
Behavioral: Physical exercises — Participants will be scheduled for supervised, regular physical training twice a week during eight weeks 8

SUMMARY:
Background:

This study is based on an innovative stepped-care protocol for the management of musculoskeletal pain in primary care, which is evaluated in a RCT. The intervention have two core features: it is theory-driven and include systematic tailoring of treatment content. The tailoring is based on a combination of empirically supported behavioural and medical determinants of pain-related disability and patients' individual perceptions on personal goals, facilitators and barriers for health behavior change. In this application, the intervention is labelled tailored behavioural medicine intervention (TBM).

Objectives:

The aim is to compare effects and cost-effectiveness of a stepped care model including advice and tailored behavioral medicine pain treatment (experimental condition) with a stepped care model including advice and physical exercises (comparison condition) for patients with low back and neck pain and/or widespread pain including fibromyalgia in primary care. A further aim is to characterize patients who benefit/do not benefit from the respective steps i.e. treatments varying in dose and content.

Methods:

A stratified randomized stepped care design is applied. Stratification is based on primary care center and patient risk profile. A consecutive selection is performed at primary care centers in southern, central and northern Sweden. According to power analysis, 364 participants should be recruited to allow for sub-group analyses. After having received a minimal intervention (step 1) comprising 'stay-active advice', participants scoring >90 on the Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) are randomly allocated to an eight-week treatment in step 2. The experimental condition includes supervised physical exercises integrated with either (a) graded activity, or (b) hierarchical graded exposure depending on risk profile, i.e. absence or presence of pain catastrophizing and fear-avoidance beliefs. The comparison condition includes supervised physical exercises irrespective of risk profile. Primary outcome is pain-related disability complemented with a comprehensive set of secondary outcomes adhering to the IMMPACT recommendations. Assessments will be made by personnel blinded for treatment condition at baseline, after step 1 and 2 respectively, and at 12- and 24-month follow-ups.

DETAILED DESCRIPTION:
STEP-UP: An innovative stepped-care model for tailored behavioral medicine treatment in the management of musculoskeletal pain in primary care

Background:

Multimodal rehabilitation and tailored behavioral medicine treatments should be provided to patients suffering from persistent and activity limiting pain according to current state-of-science. There is also evidence that a simple and specific 'stay-active advice' can produce effects comparable to effects of comprehensive treatment packages. Nevertheless, there is a gap of knowledge regarding which individuals who benefit the most from which modalities of pain treatment, at what time point, and with the highest cost-effectiveness. Accordingly, we have set up an innovative stepped-care protocol for the management of musculoskeletal pain in primary care, which is evaluated in a randomized controlled trial. The intervention have two core features: it is theory-driven and include systematic tailoring of treatment content. The tailoring is based on a combination of empirically supported behavioural and medical determinants of pain-related disability and patients' individual perceptions on personal goals, facilitators and barriers for HBC. In this application, the intervention is labelled tailored behavioural medicine intervention (TBM).

Main objectives

1. To compare the short- (post-treatment) and long-term effects (12 and 24 months follow-ups) of TBM and physical exercise treatment on everyday life activity, health related quality of life, pain severity, and sick leave (main analysis).
2. To study whether TBM tailored according to any of two pre-defined patient risk profiles: "the catastrophising/fear-avoidance profile" and "the moderate to high disability profile" are more effective compared to physical exercise treatment (sub- group analysis).
3. To characterize patients who benefit/do not benefit from (1) a minimal intervention including advice, (2) TBM and physical exercise treatment respectively
4. To identify potential moderators (e.g. pain duration, sex, outcome expectations) and mediators (e.g. catastrophising, fear of movement, self-efficacy) of treatment effects.
5. To study the cost-effectiveness within the experimental trial i.e. for the TBM versus the physical exercise treatment over the entire study period (up to 24-month follow- up).

Methods:

A stratified randomized stepped care design is applied. Stratification is based on primary care center and patient risk profile. A consecutive selection is performed at primary care centers in southern, central and northern Sweden. According to power analysis, 364 participants should be recruited to allow for sub-group analyses. After having received a minimal intervention (step 1) comprising 'stay-active advice', participants scoring >90 on the Örebro Musculoskeletal Pain Questionnaire (ÖMPQ) are randomly allocated to an eight-week treatment in step 2. The experimental condition includes supervised physical exercises integrated with either (a) graded activity, or (b) hierarchical graded exposure depending on risk profile, i.e. absence or presence of pain catastrophizing and fear-avoidance beliefs. The comparison condition includes supervised physical exercises irrespective of risk profile. Primary outcome is pain-related disability complemented with a comprehensive set of secondary outcomes adhering to the IMMPACT recommendations. Assessments will be made by personnel blinded for treatment condition at baseline, after step 1 and 2 respectively, and at 12- and 24-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* musculoskeletal pain from the low back, neck or with widespread locations

Exclusion Criteria:

* patients scoring high on the Montgomery Åsberg Depression Rating Scale (MADRS; > 35 or > 4 on the suicidal risk item)
* patients suffering from other psychiatric or severe medical co-morbidity (e.g. cancer)
* patients presenting a history and physical symptoms indicating serious spinal pathology (red flags) implying further diagnostic examination or acute measures.
* patients not being able to read, write and discuss their everyday life situation in Swedish or accepting an interpreter are not included
* patients who have completed multimodal treatments due to the current pain condition during the past two years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in pain-related disability including pain severity | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  Pain Disability Index The Chronic Pain Grade The Patient Priority Goal Questionnaire (Patient-specific measure for the study of clinical significance and goal attainment)

SECONDARY OUTCOMES:
Health related quality of life | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  SF-36
General health perceptions | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  EQ5D
Sick-absence and disability pension | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  patients self-reports of shorter sick-leave (sick-leave under 14 days), and sick-leave data collected from the Swedish Social Insurance Administration after permission from the Data Inspectorate
Pain intensity | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  Numerical rating scale (0-10), maximum, minimum average pain during past two weeks
Participants´rating of global improvement and satisfactions with treatment | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  The Patient Global Impression of Change Scale
Physical activity | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  IPAQ, Daily physical activity log

OTHER OUTCOMES:
Sick-leave | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  patients self-reports of shorter sick-leave (sick-leave under 14 days), and sick-leave data collected from the Swedish Social Insurance Administration after permission from the Data Inspectorate
Prognostic factors | baseline, after 2 week, post-treatment, 12 months follow-up, 24 months follow-up
  Self-efficacy for functional activities (The Pain Self-Efficacy Questionnaire) Fear-avoidance beliefs (The Tampa Scale of Kinesiophobia) Catastrophising (The Pain Catastrophizing Scale) Anxiety and depression (Hospital Anxiety and Depression scale , anxiety subscale) Clinical depression (The Montgomery Åsberg Depression Rating Scale (MADRS)) Psychosocial prognostic factors (Örebro Musculoskeletal Pain Questionnaire (ÖMPC), screening for risk profiles)
Demographic and background factors | baseline
  Study specific questionnaire Life-style habits, according to the national Board of Health and Welfare Personality traits (Swedish Universities Scale of Personality)
Costs | 12 months follow-up, 24 months follow-up
  Direct costs: Cost diary (including short term sick-leave), Costs for rehabilitation and production loss will be incorporated in total COSTs Indirect COSTs: SSIA registry, Standardized price labels

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Åsenlöf, Professor, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden